CLINICAL TRIAL: NCT01706172
Title: Treatment of Temporomandibular Dysfunction With Hypertonic Dextrose Injection: A Randomised Clinical Trial of Efficacy
Brief Title: Treatment of Temporomandibular Dysfunction With Hypertonic Dextrose Injection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chisel Peak Medical Clinic (Other)
Collaborators: K. Dean Reeves, M.D. (Unknown)
Responsible Party: Principal Investigator, Dr. W Francois Louw, Clinical Instructor and Physician, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMJS
Record Dates: First submitted 2012-10-11; First posted 2012-10-15 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Temporomandibular Joint Disorders
Keywords: TMD; temporomandibular; dextrose; prolotherapy
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Glucose; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dextrose 20 % Injection (Active Comparator): Injecting 20 % Dextrose and 0.2 % lidocaine intra-articularly into the TM Joint
  Interventions: Other: Injection of 20% dextrose/ 0.2% lidocaine
- Sterile Water Injection (Active Comparator): Injection of Sterile water in 0.2 % lidocaine intra-articularly into the TM joint
  Interventions: Other: Injection of 1 ml of 0.8 Sterile water /0.2% lidocaine

INTERVENTIONS:
Other: Injection of 20% dextrose/ 0.2% lidocaine — Injection at 0, 1, and 2 months of 1 ml of a solution consisting of 20% dextrose and 0.2% lidocaine.
  Arms: Dextrose 20 % Injection
Other: Injection of 1 ml of 0.8 Sterile water /0.2% lidocaine — Injection at 0, 1, and 2 months of 1 ml of a solution consisting of 0.8 sterile water and 0.2% lidocaine
  Arms: Sterile Water Injection

SUMMARY:
Dysfunction of the jaw, associated with pain in the jaw or about the jaw in the face can be quite long lasting and debilitating. Dextrose injection with a small needle has been notably helpful in preliminary studies in reducing pain and improving jaw function. This randomized trial will compare dextrose injection with sterile water injection for temporomandibular(jaw) dysfunction, also known as TMD.

DETAILED DESCRIPTION:
Longitudinal studies of subjects with temporomandibular dysfunction show a general pattern of symptom diminishment, especially in the elderly. However studies out to 2-8 years show residual symptoms in many and nearly 25% with unabated symptoms. Dextrose injection has been utilized empirically for many years and a marked reduction in pain and luxation after intra-articular and pericapsular dextrose injection has been reported in a recent RCT. However, small study size and lack of a non injection control have prevented any definitive conclusions as the additional efficacy of including dextrose in the injectate. The mechanism of action of dextrose injection was originally thought to be via a brief stimulation of the inflammatory cascade with resultant production of growth factors. However, non-inflammatory dextrose effects on growth factor production have been demonstrated, and, more recently, dextrose has been found to treat neurogenic inflammation (pain from upregulation of the TRPV1 receptor on peptidergic nerves). This has the theoretical benefit of reducing pain, regardless of the status and position of the intraarticular cartilage or degree of degenerative change of the TMD. The primary goal of this study is to evaluate the ability of dextrose injection versus saline injection to reduce pain and improve functional complaints referable to the temporomandibular joint.

ELIGIBILITY:
Inclusion Criteria:

more than 3 month history of :

* Facial Pain NRS rating > 5/10
* Jaw symptom rating > 5/10
* Jaw function issues seen on examination

Exclusion Criteria:

* Any potential acute dental issue
* Rheumatic inflammatory disease
* Chronic intake of NSAIDs or corticosteroids.
* Pain in other body location worse than jaw pain
* Pain 10/10 in other body location.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-01; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 3 months in Numerical Rating Scale (NRS) for Jaw Pain | 3 Months
  TMJ injection of 20% dextrose will result in significantly more pain relief at 3 months than injection of .2% lidocaine.

SECONDARY OUTCOMES:
Change from baseline to 3 months in Numerical Rating Scale (NRS) for Jaw Dysfunction. | 3 Months
  TMJ injection of 20% dextrose will result in significantly more improvement in Jaw Dysfunction at 3 months. Jaw dysfunction is rated based on the worst of the following: Chewing difficulty, jaw tension or stiffness, fatigue with eating, or grinding noises
TMJ injection of 20% dextrose will result in sustainable improvement in Jaw Pain to 1 year follow-up. | 1 year
  TMJ injection of 20% dextrose will result in sustainable improvement in Jaw Pain to 1 year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: W. Francois Louw, Doctor, Principal Investigator — University of British Columbia, Canada
Locations (1):
- Chisel Peak Medical Centre, Invermere, British Columbia, Canada

REFERENCES:
- [Background] Refai H, Altahhan O, Elsharkawy R. The efficacy of dextrose prolotherapy for temporomandibular joint hypermobility: a preliminary prospective, randomized, double-blind, placebo-controlled clinical trial. J Oral Maxillofac Surg. 2011 Dec;69(12):2962-70. doi: 10.1016/j.joms.2011.02.128. Epub 2011 Jul 16. PMID 21757278
- [Background] Dumais R, Benoit C, Dumais A, Babin L, Bordage R, de Arcos C, Allard J, Belanger M. Effect of regenerative injection therapy on function and pain in patients with knee osteoarthritis: a randomized crossover study. Pain Med. 2012 Aug;13(8):990-9. doi: 10.1111/j.1526-4637.2012.01422.x. Epub 2012 Jul 3. PMID 22759069
- [Background] Rabago D, Zgierska A, Fortney L, Kijowski R, Mundt M, Ryan M, Grettie J, Patterson JJ. Hypertonic dextrose injections (prolotherapy) for knee osteoarthritis: results of a single-arm uncontrolled study with 1-year follow-up. J Altern Complement Med. 2012 Apr;18(4):408-14. doi: 10.1089/acm.2011.0030. PMID 22515800
- [Background] Topol GA, Podesta LA, Reeves KD, Raya MF, Fullerton BD, Yeh HW. Hyperosmolar dextrose injection for recalcitrant Osgood-Schlatter disease. Pediatrics. 2011 Nov;128(5):e1121-8. doi: 10.1542/peds.2010-1931. Epub 2011 Oct 3. PMID 21969284
- [Derived] Louw WF, Reeves KD, Lam SKH, Cheng AL, Rabago D. Treatment of Temporomandibular Dysfunction With Hypertonic Dextrose Injection (Prolotherapy): A Randomized Controlled Trial With Long-term Partial Crossover. Mayo Clin Proc. 2019 May;94(5):820-832. doi: 10.1016/j.mayocp.2018.07.023. Epub 2019 Mar 14. PMID 30878157